CLINICAL TRIAL: NCT06043817
Title: First-In-Human Study of STX-721/PFL-721 in Participants With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Harboring EGFR or HER2 Exon 20 Insertion Mutations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STX-721-101/PFL-721CI101
Record Dates: First submitted 2023-09-01; First posted 2023-09-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer; NSCLC; EGFR/HER2 Exon 20 Insertion Mutation
Keywords: Exon 20, EGFR, HER2, NSCLC, TKI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Floors and Floorcoverings

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose Escalation (Experimental)
  Interventions: Drug: STX-721/PFL-721 (Escalated)
- Part 2: RP2D Selection (Experimental)
  Interventions: Drug: STX-721/PFL-721 (3 dose levels)
- Part 3: Dose Expansion (Experimental)
  Interventions: Drug: STX-721/PFL-721 (RP2D)

INTERVENTIONS:
Drug: STX-721/PFL-721 (Escalated) — STX-721/PFL-721 dose will be escalated per cBLRM-design.
  Arms: Part 1: Dose Escalation
Drug: STX-721/PFL-721 (3 dose levels) — Participants will receive STX-721/PFL-721 at one of three dose levels.
  Arms: Part 2: RP2D Selection
Drug: STX-721/PFL-721 (RP2D) — Participants will receive the RP2D of STX-721/PFL-721.
  Arms: Part 3: Dose Expansion

SUMMARY:
Study STX-721-101/PFL-721CI101 is an open label, Phase 1/2 study evaluating the safety, tolerability, pharmacokinetic (PK) exposure, and preliminary antitumor activity of STX-721/PFL-721 in participants with non-small cell lung cancer (NSCLC) carrying EGFR or HER2 exon 20 insertion (ex20ins) mutations.

ELIGIBILITY:
Key Inclusion Criteria:

1. Has histologically- or cytologically confirmed diagnosis of NSCLC Stage IIIB/C or IV not eligible for curative intent surgery or chemoradiation
2. Part 1: Tumor tissue EGFR or HER2 exon 20 insertion mutations confirmed by qualified local laboratories. Parts 2 and 3: EGFR/HER2 exon 20 insertion mutations confirmed by qualified local laboratories
3. Part 1: Has received all approved therapies for advanced or metastatic NSCLC or is ineligible. Part 2 and Part 3: Has received at least 1, but not more than 2, prior lines of treatment for advanced or metastatic NSCLC, 1 of which must be platinum-based chemotherapy unless contraindicated
4. Has documented tumor progression (based on radiological imaging)
5. Has new or recent tumor biopsy (collected at screening, if feasible) or archival tumor specimen collected in the past 10 years available for genomic profiling
6. Has at least one measurable tumor lesion per RECIST v1.1
7. Is ≥18 years of age at the time of signing the ICF
8. Has Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Key Exclusion Criteria:

1. Has a tumor that is known to harbor EGFR ex20ins p.H773_V774insH variant, or any EGFR kinase domain activating mutation concurrent with either a T790M and/or C797S resistance mutations
2. Has history (within ≤2 years before screening) of solid tumor or hematological malignancy that is histologically distinct from NSCLC
3. Has symptomatic brain or spinal metastases
4. Has toxicities from previous anticancer therapies that have not resolved to baseline levels or to CTCAE Grade ≤1, except for alopecia and peripheral neuropathy
5. Has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., could compromise the participant's well-being) or would prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Part 1 Dose Escalation (MTD): Dose Escalation - Number of participants who experience at least 1 DLT during the first 28 days of treatment | 28 days
Part 1 Dose Escalation (OBD): Dose Escalation - Number of participants who experience at least 1 DLT during the first 28 days of treatment | 28 days
Part 2 RP2D Selection: C(max) of STX-721/PFL-721 | 1 year
Part 2 RP2D Selection: AUC(0-inf) of STX-721/PFL-721 | 1 year
Part 2 RP2D Selection: AUC(0-t) of STX-721/PFL-721 | 1 year
Part 2 RP2D Selection: AUC(0-τ) of STX-721/PFL-721 | 1 year
Part 2 RP2D Selection: Number of participants with confirmed objective response rate (ORR) defined as the percentage of participants with partial response (PR) or complete response (CR) based on RECIST v1.1 per investigator assessment. | 1 year
Part 3 Dose Expansion: Number of participants with confirmed ORR defined as the percentage of participants with PR or CR based on RECIST v1.1 per investigator assessment. | 1 year

CONTACTS AND LOCATIONS:
Locations (23):
- United States (9):
  - City of Hope, Duarte, California
  - City of Hope, Huntington Beach, California
  - City of Hope, Irvine, California
  - Levine Cancer Institute - Charlotte, Charlotte, North Carolina
  - Thomas Jefferson University Research Facility, Philadelphia, Pennsylvania
  - SCRI Oncology Partners - PPDS, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah - Huntsman Cancer Institute - PPDS, Salt Lake City, Utah
  - NEXT Virginia, Fairfax, Virginia
- France (3):
  - EDOG Institut de Cancerologie de l'Ouest - PPDS, Saint-Herblain, Loire-Atlantique
  - Institut Claudius Regaud - PPDS, Toulouse
  - Gustave Roussy, Villejuif
- Germany (2):
  - Charité - Universitätsmedizin Berlin (CBF) - Hindenburgdamm 30, Berlin
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
- Nederlands Kanker Instituut-Antoni van Leeuwenhoek Ziekenhuis, Amsterdam, Netherlands
- South Korea (2):
  - Chungbuk National University Hospital, Cheongju-si
  - CHA Bundang Medical Center, CHA University, Seongnam-si
- Spain (4):
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga, Malaga
  - Instituto de Investigacion Oncologica Vall dHebron (VHIO) - EPON, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei